CLINICAL TRIAL: NCT06477783
Title: Prospective Observational Study on the Clinical Efficacy of Teclistamab in Patients With Relapsed and Refractory Multiple Myeloma in Belgium
Brief Title: Study on the Clinical Efficacy of Teclistamab
Acronym: TECTONIC
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Other Study IDs: 64007957MMY4010
Record Dates: First submitted 2024-05-14; First posted 2024-06-27 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-03

CONDITIONS: Multiple Myeloma; Hematologic Diseases
Keywords: Teclistamab; Tecvayli; Hematology; Efficacy; Safety
MeSH Terms: conditions — Multiple Myeloma; Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Relapsed or refractory multiple myeloma patients: Patients aged 18 years or older diagnosed with relapsed or refractory multiple myeloma, who received at least 3 prior lines of treatment. They should be refractory to at least 1 proteasome inhibitor, at least 1 immunomodulatory agent, and an anti-CD38 monoclonal antibody. After confirmation of disease progression, the patients will start treatment with teclistamab per routine clinical care or will have started with teclistamab treatment ≤14 days before intended screening visit
  Interventions: Drug: Teclistamab

INTERVENTIONS:
Drug: Teclistamab — Intervention is part of standard clinical care, as Tecvayli/Teclistamab is reimbursed for this group of patients.
  Other Names: Tecvayli

SUMMARY:
The aim of this study is to assess the clinical efficacy and safety of the anti-BCMA/CD3 bispecific antibody teclistamab (Tecvayli®) in a prospective, real-life setting in Belgium.

DETAILED DESCRIPTION:
To assess the clinical efficacy and safety of teclistamab (Tecvayli®) in relapsed/refractory multiple myeloma patients who have received at least 3 prior lines of treatment and who will receive teclistamab (Tecvayli®) as the next treatment. Patients will be followed up prospectively until the end of study (24 months/2 years), or until disease progression, withdrawal of consent death or loss to follow-up, whichever occurs first. Each patient will have a monthly follow-up from baseline until 6 months of treatment with teclistamab. Then, data will be collected every 3 months until the end of study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Written informed consent
* Has a diagnosis of relapsed and refractory multiple myeloma
* Has already received at least three previous treatments
* Is refractory to at least 1 proteasome inhibitor, at least 1 immunomodulatory agent, and an anti-CD38 monoclonal antibody
* Evidence of disease progression on the last line of therapy, based on determination of response by the IMWG response criteria
* Anticipated to start treatment with teclistamab per routine clinical care or has started with teclistamab treatment ≤14 days before intended screening visit

Exclusion Criteria:

* Has participated in a teclistamab trial (teclistamab or control arm) or teclistamab Single Patient Request (SPR) program
* Has started teclistamab treatment >14 days before intended screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients with relapsed or refractory multiple myelome who will be treated with teclistamab (Tecvayli®)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | At baseline, monthly until end of study (maximum 24 months)
  The primary objective is the overall response rate (partial response (PR) or better) according to the 2016 IMWG response criteria of Multiple myeloma.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | At baseline, monthly until end of study (maximum 24 months)
  The length of time during and after the treatment during which a patient lives with the disease but it does not get worse.
Overall survival (OS) | At baseline, monthly until end of study (maximum 24 months)
  Duration of time between start of the treatment and up to the time of death.
Incidence of (serious) adverse events | At baseline, monthly until end of study (maximum 24 months)
  Incidence and severity of (serious) adverse events with with focus on hematological AE's (≥ grade 3), cytokine release syndrome (CRS) rate, Immune effector cell-associated neurotoxicity syndrome (ICANS) and infections (≥ grade 2) and serious adverse events related to teclistamab (Tecvayli®).
Depth of response | At baseline, monthly until end of study (maximum 24 months)
  Evaluation of response in terms of depth. Assessment of response according to the 2016 IMWG response criteria of Multiple myeloma.
Time to response (TTR) | At baseline, monthly until end of study (maximum 24 months)
  Assessment of the time it takes for a patient to achieve partial response (PR) or better.
Duration of response | At baseline, monthly until end of study (maximum 24 months)
  Assessment of the length of time during which a patient experiences a partial response (PR) or better. It is measure from the start of treatment until disease progression or death.
Minimal Residual Disease (MRD) assessment | At suspected CR, every 6 months thereafter until end of study (maximum 24 months)
  Evaluation of treatment efficacy by monitoring for the presence of a small number of cancer cells that are left in the body. MRD assessment will be done with Next Gen Flow (NGF) or Next Gen Sequencing (NGS).
Time to next treatment (TTNT) | At baseline, monthly until end of study (maximum 24 months)
  Assessment of the time interval between initiation of treatment with Tecvayli® and commencement of the next line of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Delforge, MD, PhD, Principal Investigator — UZ Leuven Gasthuisberg
Locations (17):
- Belgium (17):
  - Imelda, Bonheiden, Antwerpen
  - Universitair Ziekenhuis Antwerpen (UZA), Edegem, Antwerpen
  - Grand Hôpital de Charleroi, Charleroi, Henegouwen
  - EpiCURA, Hornu, Henegouwen
  - CHU Ambroise Paré, Mons, Henegouwen
  - Jessa Ziekenhuis, Hasselt, Limburg
  - CHR Citadelle, Liège, Liège
  - CHU Liège, Liège, Liège
  - CHU UCL Namur, Yvoir, Namur
  - Algemeen Ziekenhuis Maria Middelares (AZMM), Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Gent (UZ Gent), Ghent, Oost-Vlaanderen
  - Vitaz, Sint-Niklaas, Oost-Vlaanderen
  - Institut Jules Bordet, Brussels, Vlaams-Brabant
  - UCL Saint Luc, Brussels, Vlaams-Brabant
  - AZ Groeninge, Kortrijk, West-Vlaanderen
  - AZ Delta, Roeselare, West-Vlaanderen
  - UZ Leuven Gasthuisberg, Leuven

IPD SHARING:
Plan to Share IPD: No